CLINICAL TRIAL: NCT02893644
Title: Optical Coherence Pachymetry (OCP) to Evaluate Central Corneal Ablation Depth in Myopic Femtosecond Laser in Situ Keratomileusis (LASIK)
Brief Title: Optical Coherence Pachymetry to Evaluate Central Corneal Ablation Depth in Myopic Femtosecond Laser in Situ Keratomileusis
Acronym: PACO
Status: Completed | Type: Observational
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Other Study IDs: JFO_2013-15
Record Dates: First submitted 2016-08-30; First posted 2016-09-08 (Estimated); Last update posted 2017-03-20 (Actual); Status verified 2017-03

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective

SUMMARY:
Prospective study aiming to measure central ablation depth during excimer laser surgery in myopic patients operated with femtosecond laser assisted LASIK with intraoperative OCP, before and after laser ablation. This measurement will be compared with pre and 1 month postoperative topography differential pachymetric measurements.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years old
* undergoing refractive surgery with LASIK
* with myopic or compound myopic astigmatism ametropia
* without irregular cornea and topographical sign of keratoconus
* preoperative corneal thickness compatible with LASIK

Exclusion Criteria:

* hyperopia
* opposition to participate in the study
* no health insurance coverage
* patient under legal protection
* pregnant or breastfeeding patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients undergoing refractive surgery with LASIK
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2014-05-26 (Actual); Primary Completion 2016-07-26 (Actual); Study Completion 2017-03-15 (Actual)

PRIMARY OUTCOMES:
depth of central corneal ablation | 1 month after surgery
  measured in microns with OCP

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Luc FEBBRARO, MD, Principal Investigator — Fondation OPH A de Rothschild
Locations (1):
- SALOMON, Paris, France